CLINICAL TRIAL: NCT01029444
Title: Effects of Pulsatile Intravenous Insulin on Brittle Diabetes and Glucose Control
Brief Title: Effects of Pulsed Intravenous (IV) Insulin on Brittle and Uncontrolled Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other)
Responsible Party: Betty Tuller PhD Professor of Complex Systems and Brain Sciences, Florida Atlantic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H09-66 BUD
Record Dates: First submitted 2009-08-06; First posted 2009-12-10 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Pulsatile intravenous insulin; Oral carbohydrate loading; Respiratory Quotients; Hypoglycemia; Hyperglycemia; Diabetes Mellitus, with complications
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Diabetes Complications | interventions — Insulin, Regular, Human; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin (Experimental): Brittle diabetic patients or patients with uncontrolled blood sugars will complete blood sugar diaries weekly and have hemoglobin A1c lab tests performed quarterly to evaluate progress in stabilizing blood sugars.
  Interventions: Procedure: Pulsatile Intravenous Insulin Therapy (Humulin, Humulog, Novolog )

INTERVENTIONS:
Procedure: Pulsatile Intravenous Insulin Therapy (Humulin, Humulog, Novolog ) — Patients receive weekly treatments of Pulsatile Intravenous insulin therapy. The patient's Endocrinologist determines the insulin dosage each week based upon the patient's response to treatment RQ levels and their insulin resistance.

SUMMARY:
The purpose of this study is to determine if restoring normal metabolic function in patients with either type I or type II diabetes can improve the impact of the consequences of diabetic complications specifically on the wide swings in blood glucoses with erratic control even under optimal conditions. Patients are treated once a week with pulsatile intravenous insulin therapy mimicking normal insulin secretion. Blood sugar diaries and laboratory tests including quarterly Hemoglobin A1c levels are monitored to measure progress and outcomes.

DETAILED DESCRIPTION:
It is known that the glucose metabolic pathway (glycolysis) is the primary fuel generator in the brain and nerve tissue, the heart and vascular tissue, the eye, the kidney and the liver Deficient metabolic states such as seen in the glucose metabolism of diabetics can lead to sequelae. These damaging effects are exacerbated by altered cellular metabolites, specifically the increase in catabolic and decrease in anabolic factors. It has been shown over the past twenty years that normalization of metabolism in diabetic patients can be accomplished by mimicking the normal endogenous insulin pattern (i.e., in pulses). Pulsatile intravenous insulin infusion has been demonstrated to stabilize the erratic wide swings in blood glucose levels and the overall stabilization of hyperglycemic and hypoglycemic events in Type 1 diabetic patients. This study was established to evaluate the effect of providing pulsatile intravenous insulin therapy on both type 1 and type 2 diabetes to determine the effect on improving diabetic control on patients with high blood glucose levels in spite of multiple insulin injections and wide swings in blood sugar despite good control.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 30 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQ's higher than 1.05. The RQ can be followed serially and this is done before and after each pulsatile IV insulin treatment, during the 3 successive sessions on a single treatment day. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous session.pulsatile IV insulin therapy encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those found in non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/ VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions.Patient is evaluated post session and discharged when stable.

Frequent monitoring of RQ is necessary as these levels change rapidly, depending on the fuel being utilized by the body. Pulsatile IV insulin therapy shifts metabolism from primarily fatty acid metabolism to primarily glucose metabolism. This shift is reflected by the increase in respiratory quotient. However during rest periods the RQ may fall back to lower levels. Therefore RQ's are done at the beginning and at the end of each insulin infusion session of 1 hour in order to appropriately monitor and adjust insulin and carbohydrate loads to reach optimal activation in each session

ELIGIBILITY:
Inclusion Criteria:

* The researchers will include up to 300 patients both male and female between the ages of 18 and 85 diagnosed with type 1 or type 2 diabetes mellitus.
* Self reporting or diagnosed with significant complications resulting from diabetes.
* Taking oral agents and/or insulin for diabetic control.
* Under an Endocrinologists supervision for their diabetes management.
* Endocrinologist must assess and approve patient for participation in this study.
* Ability to swallow without difficulty.
* Ability to commit to the weekly time requirements associated with the study.

Exclusion Criteria:

* Other causes of complications not related to diabetes.
* Lack of intravenous access.
* Pregnancy.
* Alcohol abuse, drug addiction or the use of illegal drugs.
* Positive HIV.
* Inability to breathe into machine for respiratory quotients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of Pulsed IV Insulin Therapy on the stabilization of blood glucose levels on patients with brittle or uncontrolled diabetes | Blood sugar diaries are collected weekly and HA1c labs are collected at baseline and quarterly to assess progress

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, PhD, Study Director — Florida Atlantic University
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States